CLINICAL TRIAL: NCT02818660
Title: Mass Spectrometry Based Cutoffs for Cortisol and 17-hydroxy-progesterone (17-OH-progesterone) After Stimulation Tests for Primary and Secondary Adrenal Insufficiency.
Brief Title: Mass Spectrometry Based Cutoffs for Cortisol After Stimulation Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/174
Record Dates: First submitted 2016-06-14; First posted 2016-06-30 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Cosyntropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Synacthen (Experimental): The patient get Synacthen to stimulate the adrenals to produce cortisol
  Interventions: Drug: Synachten

INTERVENTIONS:
Drug: Synachten — To stimulate the adrenals to increase the cortisol Production as much as possible
  Other Names: tetracosactide

SUMMARY:
There are two main stimulation tests used to decide if a patient has cortisol deficiency. It is the "synacthen test", were we stimulate the patient with intramuscular or intravenous synacthen ( ACTH) to see how much cortisol the adrenals are capable of producing, and it is the "Insulin hypoglycemia test" were we give the patient insulin to provoke a hypoglycemia, and look at the adrenal response to that stimulus. The cut off values for a normal response is based on old immunological assays no longer in use. Assays with a lot of interference and cross reactivity leading to measurement of higher values for cortisol than what we measure on the highly specific LCMS/MS ( Liquid chromatography mass spectrometry methode) that we are using for cortisol today. So, there is a need for new cut off values for a normal response to such tests. The purpose of this study is to produce such new cutoff values by performing the test in 120 healthy controls. We also want to perform the test in patient groups normally going trough this tests according to the same protocol as the control persons, to evaluate the new cutoffs in different patient groups.

DETAILED DESCRIPTION:
120 healthy controls will perform an intravenous synacthen test in our out patient clinic. We register anthropometric data, and take basal blood screening to assure they are healthy. We take basal blood and saliva samples right before start of the test ( called 0-samples). Then they get intravenous synacthen, and we take new samples at 30 minutes and 60 minutes. They are observed during the procedure. We will then calculate a new cut off value for cortisol after the test, based on the 2.5 percentile for cortisol in this population. We will also calculate the same for 17-OH-progesterone, a parameter we also look at after synacthen test in som patient groups ( patients with hirsutism, who are suspicious of having an enzyme defect in the cortisol synthesis cascade). The saliva samples will also be analyzed for cortisol and 17-OH-progesterone, to evaluate if it is possible to use saliva instead of blood samples in synacthen tests in the future. The advantage of using saliva samples is that they can be used also in patients with elevated amount of cortisol binding globulin (CBG), because it measure the free hormone that is biological active ( not both the free and the protein bound, as we measure in serum samples). This is important in patients on estrogens , and in pregnant women, that have large amount of CBG.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals not using any corticosteroids .
* Patients with clinical suspicion of primary or secondary adrenal insufficiency. -Patient suspicious of having an enzyme defect ( 21 hydroxylase deficiency) giving hirsutism.

Exclusion Criteria:

-Use of corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-05-21 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Define a cutoff level for serum cortisol after stimulation with synacthen or hypoglycemia in healthy control persons. | 2 year
  s-cortisol

SECONDARY OUTCOMES:
Define a cutoff level for serum 17-OH-progesterone after stimulation with synacthen or hypoglycemia in healthy control persons. | 2 year
  s-17-OH-progesterone
Define a cutoff level for saliva cortisol after stimulation with synacthen or hypoglycemia in healthy control persons. | 2 year
  saliva cortisol
Define a cutoff level for saliva 17-OH-progesterone after stimulation with synacthen or hypoglycemia in healthy control persons. | 2 year
  saliva 17-OH-progesterone

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Åstrøm Ueland, MD, Principal Investigator — Haukeland University Hopsital
Locations (1):
- Haukeland University hopsital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ueland GA, Methlie P, Oksnes M, Thordarson HB, Sagen J, Kellmann R, Mellgren G, Raeder M, Dahlqvist P, Dahl SR, Thorsby PM, Lovas K, Husebye ES. The Short Cosyntropin Test Revisited: New Normal Reference Range Using LC-MS/MS. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1696-1703. doi: 10.1210/jc.2017-02602. PMID 29452421
- [Result] Ueland GA, Dahl SR, Methlie P, Hessen S, Husebye ES, Thorsby PM. Adrenal steroid profiling as a diagnostic tool to differentiate polycystic ovary syndrome from nonclassic congenital adrenal hyperplasia: pinpointing easy screening possibilities and normal cutoff levels using liquid chromatography tandem mass spectrometry. Fertil Steril. 2022 Aug;118(2):384-391. doi: 10.1016/j.fertnstert.2022.05.012. Epub 2022 Jun 18. PMID 35725670